CLINICAL TRIAL: NCT04679870
Title: An Open-label, Phase IIa Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral GB2064 (a LOXL2 Inhibitor) in Participants With Myelofibrosis (MF)
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral GB2064 in Participants With Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Galecto Biotech AB (Industry)
Collaborators: OPIS s.r.l (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYLOX-1; 2020-003087-45 (EudraCT Number)
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Myelofibrosis
Keywords: GB2064; Myelofibrosis; LOXL-2; PAT1251
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: All subjects eligible for the study will receive GB2064 1000mg, twice a day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GB2064 (Experimental): GB2064 will be administered orally as 4 x 250 mg tablets twice a day.
  Interventions: Drug: GB2064

INTERVENTIONS:
Drug: GB2064 — GB2064 (formerly PAT-1251) is a high-affinity, selective, mechanism-based, small molecule inhibitor of LOXL2, administered twice a day

SUMMARY:
This study is an open label, phase IIa trial in subjects with Myelofibrosis

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of orally administered GB2064 a LOXL-2 inhibitor over 9 months. Subjects will receive doses of GB2064, given twice per day to participants with primary or secondary Myelofibrosis

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy all of the following criteria at the Screening visit:

1. Adult male or female participants ≥ 18 years of age at enrolment:

   1. Female participants may be of non-childbearing potential defined as permanently sterile or postmenopausal, or female participants considered to be of childbearing potential who agree to use highly effective birth control methods until 90 days after the follow-up visit. Female participants should refrain from ova donation from the date of Enrolment (Day -1) until 90 days after the follow-up visit.
   2. Male participants will agree to use contraception throughout the study and until 90-days after the Follow-up visit. Male participants must agree to refrain from sperm donation from the date of Enrolment (Day -1) until 90 days after the follow-up visit.
2. Diagnosis of PMF or SMF with intermediate -2 or high-risk disease according to the Dynamic International Prognostic Scoring System (DIPSS)-plus or if with low risk disease then with symptomatic splenomegaly as defined by sonographic assessment as spleen length of >12 cm or by physical examination as ≥ 5 cm below left costal margin.
3. Participants who are not currently taking a Janus kinase (JAK) inhibitor (e.g. ruxolitinib or fedratinib) and are therefore refractory, intolerant or ineligible for a JAK inhibitor according to appropriate guidelines (including local guidelines).
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Required baseline laboratory status:

   1. Absolute platelet count (APC) ≥ 50 x 109/L
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (1500/mm3)
   3. Serum direct bilirubin ≤ 2.0 x ULN (upper limit of normal)
   4. AST (SGOT) or ALT (SGPT) [if both measured, then this applies to both measurements] ≤ 2.5 x ULN, except for participants with MF involvement of the liver who must have levels ≤ 5 x ULN
   5. Estimated Glomerular Filtration Rate (eGFR) or creatinine clearance (CrCl) (CrCl calculated by the Cockroft and Gault method) ≥ 30 ml/min/1.73 m2.
   6. Peripheral blood blasts <10%
6. Treatment-related toxicities from prior therapies must have resolved to Common Terminology Criteria for Adverse Events (CTCAE) Grade ≤ 1.
7. Participants must have a documented history of transfusion records (if there have been any such transfusions) in the preceding 12 weeks to Day 1.

Exclusion Criteria:

1. Current treatment with a JAK inhibitor (e.g. ruxolitinib or fedratinib) or a history of treatment with a JAK inhibitor within two weeks of enrolment.
2. Positive hepatitis panel and/or positive HIV test.
3. Any concurrent severe and/or uncontrolled medical conditions that could increase the participant's risk for toxicity while in the study or that could confound discrimination between disease- and study treatment-related toxicities. Any planned major surgery during the study period
4. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   1. History or presence of ventricular tachyarrhythmia.
   2. Presence of unstable atrial fibrillation (ventricular response > 100 bpm); Participants with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria.
   3. Clinically significant resting bradycardia (< 50 bpm) and use of a cardiac pacemaker or implantable cardioverter defibrillator.
   4. Angina pectoris or acute myocardial infarction ≤ 90 days prior to starting study drug.
   5. Other clinically significant heart disease (e.g., symptomatic congestive heart failure; uncontrolled arrhythmia or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen).
5. Participants who are currently receiving chronic (> 14 days) treatment with corticosteroids at a dose > 10 mg of prednisone (or its glucocorticoid equivalent) per day, or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug.
6. Participants with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of GB2064 as per physician's opinion.
7. Participants who received radiotherapy within the last month prior to screening procedures, or patients who received splenectomy in the previous three months or are scheduled for the procedure in the next three months.
8. Participants who had a history of malignancy in the past 3 years, except for treated early stage squamous, basal cell carcinoma or treated, localised prostate cancer.
9. Presence of clinically meaningful active bacterial, fungal, parasitic or viral infection which requires therapy.
10. Previous history of Progressive Multifocal Leuko-encephalopathy (PML).
11. Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive β- HCG laboratory test.
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 90 days after study treatment. Highly effective contraception methods must be used.
13. Sexually active males must use a condom during intercourse while taking the drug and for 90 days after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
14. Hypersensitivity to GB2064 and/or its excipients.
15. Participants unable or unwilling to comply with protocol requirements.
16. Participants related to PI/site staff.
17. Participants who have had a hematopoietic stem cell transplantation.
18. Participants who are eligible, have a donor and are willing to undergo a hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of GB2064: AE | 9 Months
  Incidence and severity of adverse events as reported by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Schlenk, MD, Principal Investigator — Universitätsklinikum Heidelberg, Germany
Locations (11):
- MD Andersson Cancer Hospital, Houston, Texas, United States
- Woden Dermatology, Canberra, Australia
- Germany (4):
  - Heinrich-Heine-University Dusseldorf, Düsseldorf
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universität Leipzig, Leipzig
  - Klinikum rechts der Isar der Technischen Universitaet Munchen, München
- Italy (5):
  - University of Bologna Sant Orsola Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga di Orbassano, Orbassano
  - Azienda Socio-Sanitaria Territoriale dei Sette Laghi, Varese

IPD SHARING:
Plan to Share IPD: No